CLINICAL TRIAL: NCT01532817
Title: Non-Invasive Neurostimulation of the Vagus Nerve With the AlphaCore™ Device, for the Relief of Acute Bronchoconstriction Due to Asthma
Brief Title: Relief of Acute Bronchoconstriction/Asthma Using the Non-Invasive AlphaCore Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ElectroCore INC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BC-US-06
Record Dates: First submitted 2012-02-10; First posted 2012-02-15 (Estimated); Results first posted 2018-04-09 (Actual); Last update posted 2018-04-09 (Actual); Status verified 2018-04

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- alphacore (Experimental): noninvasive neurostimulation of the vagus nerve
  Interventions: Device: AlphaCore

INTERVENTIONS:
Device: AlphaCore — A single 90 second stimulation to the vagus nerve on the right side of the neck

SUMMARY:
The purpose of this pilot study is to collect preliminary clinical data related to the safety and preliminary clinical benefits of non-invasive vagal nerve stimulation with the AlphaCore™ device for the relief of acute bronchoconstriction due to asthma.

Up to 30 subjects who meet all inclusion/exclusion criteria and consent to participate in the study may be enrolled at up to 5 investigational (study) sites. The study sites are clinic settings capable of treating any potential complications of bronchoconstriction, an acute exacerbation of asthma, and any emergencies associated with use of the investigational device.

DETAILED DESCRIPTION:
Subjects will be screened, consented and enrolled at the first visit. Subjects will return to the second visit where they are experiencing shortness of breath and will be treated with the alphacore. Breathing and vital signs will be measured before, during and after the stimulation. The study is concluded on the third visit, 7 days later.

ELIGIBILITY:
INCLUSION CRITERIA: VISIT 1

1. Is able to give written Informed Consent.
2. Is between the ages of 18 and 65 years, male or female.
3. Has a known history of mild to moderate asthma for at least 1 year as defined by GINA Guidelines.
4. Is using a short acting beta-agonist for relief/rescue of asthma..
5. At Visit 1, demonstrates current or historical (within 1 year) FEV1 reversibility of at least 12% (and 200ml) or greater within 15-30 minutes following administration of 4 inhalations of albuterol.

EXCLUSION CRITERIA: VISIT 1

1. Has a history of lung cancer, chronic obstructive pulmonary disease (COPD), or other co-morbidity associated with irreversible narrowing of the airways.
2. Has an abscess or other infection or lesion (including lymphadenopathy) at the AlphaCore™ treatment site.
3. Has known or suspected moderate to severe atherosclerotic cardiovascular disease, carotid artery disease (e.g. bruits or history of TIA or CVA) or congestive heart failure (CHF).
4. Has suspected or confirmed sepsis.
5. Has a clinically significant irregular heart rate or rhythm.
6. Has experienced recent clinically significant changes in blood pressure, has uncontrolled high blood pressure, or is presently receiving pressors to maintain blood pressure.
7. Is currently implanted with an electrical and/or neurostimulator device, including but not limited to cardiac pacemaker, defibrillator, vagal neurostimulator, deep brain stimulator, spinal stimulator, bone growth stimulator, or cochlear implant.
8. Has a history of carotid endarterectomy or vascular neck surgery on the right side.
9. Has been implanted with metal cervical spine hardware.
10. Has a recent or repeated history of syncope.
11. Has a recent or repeated history of seizures.
12. Is pregnant or nursing, or of childbearing years and is unwilling to use an accepted form of birth control.
13. Is participating in any other therapeutic clinical investigation or has participated in a clinical trial in the preceding 30 days.
14. Belongs to a vulnerable population or has any condition such that his or her ability to provide informed consent, comply with follow-up requirements, or provide self-assessments is compromised (e.g., homeless, developmentally disabled, prisoner).
15. Is a relative of or an employee of the Investigator or the clinical study site.

INCLUSION CRITERIA: VISIT 2

1. No changes have occurred in the patient's health or status relative to the original inclusion and exclusion criteria and the patient continues to be eligible for participation in the study.
2. Either (i) develops subjective symptoms of asthma (wheezing, shortness of breath, cough) for which the patient would normally self-medicate with a short acting beta agonist, and/or (ii) documents a drop of 20% from screening PEF scores as recorded in their patient diary.
3. At Visit 2, FEV1 is the same or lower than the screening FEV1 previously measured at visit 1 or the PEF is the same or lower than the screening previously measured at Visit 1.

EXCLUSION CRITERIA: VISIT 2

1. The patient self-administered a short-acting beta agonist within 6 hours prior to onset of asthma symptoms.
2. The patient induced an asthma exacerbation by withholding their pre-treatment medication used for exercise-induced bronchoconstriction (EIB).
3. Has signs and symptoms of asthma instability at Visit 2:

   * Lung Function: FEV1 < 50 % predicted.
   * Signs and symptoms of extreme respiratory distress at rest.
   * Rapid deterioration in respiratory status (sudden change in respiratory rate, decrease in oxygen saturation, change in consciousness, etc.).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Erico, Study Chair — ElectroCore INC
Locations (3):
- United States (3):
  - Allergy and Asthma, San Diego, California
  - CRI, Minneapolis, Minnesota
  - Vital Prospects Clinical Research Institute, Tulsa, Oklahoma

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Alphacore
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Open label 30 patient population
Arm/Group | Alphacore
Number analyzed (Participants) | 30
Age, Customized [Median (Full Range); unit: years]
  Age | 30 [20 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 17
  Black | 8
  Hispanic | 4
  Other | 1
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Safety- Number of Participants With Adverse Events
Description: Safety- number of participants with adverse events, including device-related, serious or unanticipated
Time Frame: From time subject signs the consent through the 1-week follow-up visit
Population: Open label study 30 participants
Measure: Count of Participants; unit: Participants
Arm/Group | Alphacore
Number analyzed (Participants) | 30
Participants | 10

ADVERSE EVENTS:
Time Frame: From screening visit 1 to visit 3 follow up, 9 weeks.
Arm/Group | Alphacore
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 10/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alphacore (N=30)
Local site neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Increased chest congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sensation of muscle tightness/spasm from right ear to right wrist (Musculoskeletal and connective tissue disorders) | 1 (1)
Increased mucus in post oropharynx (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Faint localised area of erythema on anterior biceps bilaterally (Skin and subcutaneous tissue disorders) | 1 (1)
Allergic reaction to food (Immune system disorders) | 1 (1)
Upper body jitteriness (Nervous system disorders) | 1 (1)
Sensation of musculoskeletal tenseness/tightness through upper body (Musculoskeletal and connective tissue disorders) | 1 (1)
Right neck skin itching (Skin and subcutaneous tissue disorders) | 1 (1)
Tingling sensation on right side of neck (Nervous system disorders) | 1 (1)
Torticollis muscular (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Viral respiratory syndrome (Infections and infestations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less